CLINICAL TRIAL: NCT06930768
Title: Evaluation of the Efficacy of NeoThelium FT in the Healing of Venous Leg Ulcers: A Randomized Controlled Multicenter Trial
Brief Title: Evaluating the Efficacy of NeoThelium FT in the Treatment of Venous Leg Ulcers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuScience Medical Biologics, LLC (Industry)
Collaborators: SygNola, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VELOCITY
Record Dates: First submitted 2025-04-01; First posted 2025-04-16 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Venous Leg Ulcer
Keywords: Chronic wounds; Wound Medicine; Cellular, Acellular, Matrix-like Product (CAMP); Cellular and/or Tissue Product (CTP); Dehydrated Complete Human Placental Membrane (dCHPM)
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The subject will be randomized to one of the following treatments:
  * Standard of care
  * NeoThelium FT in addition to standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Standard of Care (Active Comparator): Wound cleansing, Sharps debridement, Dressing for moisture balance, Offloading
  Interventions: Other: Standard of Care
- Intervention: NeoThelium FT & Standard of Care (Experimental): Wound cleansing, sharps debridement, NeoThelium FT application, Dressing for moisture balance, Offloading
  Interventions: Other: NeoThelium FT

INTERVENTIONS:
Other: Standard of Care — Wound cleansing, Sharps debridement, Dressing for moisture balance, Offloading
  Arms: No Intervention: Standard of Care
Other: NeoThelium FT — NeoThelium FT is a dehydrated wound covering derived from donated human placental tissue. NeoThelium FT is a dual-layer membrane with amnion and chorion combination layers.
  Arms: Intervention: NeoThelium FT & Standard of Care

SUMMARY:
This is a randomized controlled trial evaluating the efficacy of NeoThelium FT in conjunction with standard of care vs. standard of care alone in treating venous leg ulcers.

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will be randomly assigned to one of two groups: either standard of care alone, or standard of care plus NeoThelium FT. As this is a post-marketing study, it will gather information about how effective the treatment is in treating venous leg ulcers. All subjects will complete two week screening phase prior to being randomized into a treatment arm. Treatment arms will consist of NeoThelium FT in conjunction with standard of care, vs. standard of care alone. The primary endpoint will be the percentage of target ulcers that achieve complete wound closure within 16 weeks. Secondary endpoints consist of wound area reduction rates, time to closure, follow-up closure, and pain assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of Venous Insufficiency with an open wound to the lower extremity
3. Subject has a Venous Leg Ulcer present for 4 weeks or greater (documented in medical record), and less than 12 months duration if being treated with continuous SOC
4. Subject has a Venous Leg Ulcer with a historical wound measurement showing less than 50% healing in 30 days prior to randomization
5. Subject has a Venous Leg Ulcer with screening wound measurement showing less than 25% healing in 14 days prior to randomization
6. Subject has a Venous Leg Ulcer Wagner 1, 2, and 3 without infection or clinically visible exposed bone
7. Index ulcer is a minimum of 1cm2 and a maximum of 40cm2 at first treatment visit
8. Venous Leg Ulcer is being treated with compression therapy for 14 days prior to randomization
9. Adequate circulation of ulcer demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to randomization
10. Index ulcer is free of infection prior to randomization and during screening phase noted with the NERDS Assessment. Infection must be adequately treated and controlled prior to randomization.
11. Index ulcer is free of necrotic debris prior to NeoThelium FT application
12. Female subjects of childbearing potential having a negative pregnancy test prior to randomization
13. Subject is able and willing to follow the protocol requirements
14. Subject had signed informed consent
15. If 2 or more ulcers are present, the ulcers must be separated by at least 1 cm

Exclusion Criteria:

1. Subject has a known life expectancy of <1 year
2. Subject is unable to comply with protocol treatment
3. Subject has major uncontrolled medical disorders in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders that may affect wound healing
4. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound
5. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
6. Known contraindications to tissue-engineered allograft
7. Concurrent participation in alternative clinical trial that involves investigational drug or product interfering with wound treatment and/or healing
8. Wound reduces in area by ≥25% after 14 days of SOC prior to randomization
9. Subject is pregnant or breastfeeding
10. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the ulcer surface for >2 weeks duration within 30 days prior to randomization; or anticipated use of the above during the course of the study
11. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to randomization
12. Venous Leg Ulcer with active infection
13. Wound depth with visible exposed bone
14. HBOT within 14 days prior to randomization
15. Revascularization surgery on the index ulcer leg within 30 days of screening phase
16. Index ulcer suspicious of neoplasm in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-12 weeks
  The primary endpoint will be the percentage of target ulcers that achieve complete wound closure.

SECONDARY OUTCOMES:
Percentage Wound Area Change | 1-12 weeks
  The percentage change in wound area from TV-1 to TV-13 will be measured weekly using digital photographic planimetry and physical examination.
Time to Closure | 1-12 weeks
  Average number of grafts and/or weeks used to achieve wound closure
Follow-Up Closure | 2 weeks
  Number of wounds remaining closed during the 2-week follow-up
Pain Assessment | Day 0, Day 14, Day 35, Day 56, Day 84
  Change in pain associated with the target ulcer will be assessed using the Numeric Pain Rating Scale at designated time points

OTHER OUTCOMES:
Wound closure rate in comparison to initial area | Day 0 through Day 84
  Wound healing rate vs wound area categories 0.5-1 cm2, >1-3cm2, >3-5cm2, etc.
Adverse Events and Serious Adverse Events | Day -14 through 91 days
  The number and nature of adverse events (AEs) and series adverse events (SAEs) occurring during the study will be tracked and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Ferguson, DNP, Study Director — SygNola, LLC

IPD SHARING:
Plan to Share IPD: No